CLINICAL TRIAL: NCT06618456
Title: Hypnosis Induction and Height Experience in Virtual Reality - Comparison With Control Group and Investigation of the Effect of Three Sessions
Brief Title: Hypnosis Induction and Height Experience in VR - Control Group Comparison and Three Sessions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Milton Erickson Gesellschaft für klinische Hypnose (Unknown); Milton Erickson Gesellschaft Stiftung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 521/2019BO2
Record Dates: First submitted 2024-05-07; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-03

CONDITIONS: Acrophobia
Keywords: Virtual Reality; Hypnosis; Acrophobia; Exposition
MeSH Terms: conditions — Acrophobia

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of the two groups (experimental group / control group). In the experimental group participants undergo a VR-supported trance induction. The participants in the control group are the same VR-environment but do not receive a trance induction. Then there is an automatic transition to the altitude confrontation (also in VR) in both groups. The experimental group receives hypnotic suggestions via audio, that partially refer to a tree positioned next to the participants in the VR-altitude-confrontation. In the control group this tree is replaced by a parasol in the VR and the text via audio. Besides from that they receive the same text as the experimental group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants undergo an VR-supported trance induction. Participants will see an underwater world adapted to the sound (i.e. text) of the trance. The following exposure will be nearly the same for both groups (see differences in study design).
  Interventions: Behavioral: VR dive (with Hypnosis); Behavioral: Height exposure
- Control group (Active Comparator): Participants see the same underwater world in VR but receive no trance induction. The following exposure will be nearly the same for both groups (see differences in study design).
  Interventions: Behavioral: VR dive (without Hypnosis); Behavioral: Height exposure

INTERVENTIONS:
Behavioral: VR dive (with Hypnosis) — Participants experience a VR dive through a friendly underwater world. They get a trance induction via audio.
  Arms: Experimental group
Behavioral: VR dive (without Hypnosis) — Participants experience a VR dive through a friendly underwater world. They are informed that this part of the VR is a familiarization phase to the VR and they do not get a trance induction.
  Arms: Control group
Behavioral: Height exposure — The participants go through a height exposure. They start at the ground level of a virtual city and move upwards in 3 meter steps until they reach a height of 60 meters. Participants focus on a yellow spot on a balcony in front of them, so that they can recognise the depth perimeter.

SUMMARY:
This study attempts to test wether a VR-supported trance induction and a subsequent exposure to altitude in VR with hypnotic suggestions via Audio reduces acrophobia more than a control-group intervention without trance induction. Furthermore the study attempts to test if three sessions of the interventions within three weeks can lead to a stronger reduction of acrophobia than only one session.

Participants will be selected via an online survey according to their score on the Height Interpersonal Questionnaire (HIQ). At the start of the study, participants will be screened by professional clinicians for any mental disorders. In the laboratory they will undergo one of the two interventions in VR (experimental group / control group) and complete questionnaires for three times within three weeks. On a separate day within these three weeks they will be placed in a 30-minute trance to test their suggestibility.

DETAILED DESCRIPTION:
Prior to the measurement, those interested in the study will complete a screening questionnaire on acrophobia (HIQ) online. Besides they will be asked if they ever had negative experiences with VR or hypnosis. Only persons who do not report negative experiences with VR or hypnosis and who attain a HIQ score bigger than 29 will be invited to take part in the study. At the first appointment in the laboratory a screening with SCID questions about disorders that would lead to exclusion is conducted. On the basis of this second screening participants will be admitted to the study. Failure to meet the criteria (see eligibility section) will exclude participants from the study. At the start of the assessment session, participants will complete a sociodemographic questionnaire and again the HIQ.

Participants are randomly assigned to one of the two groups. Based on group affiliation they either undergo a VR-supported trance induction or the same VR-program without the trance induction. Then there is an automatic transition to the altitude confrontation. Both groups receive the same VR altitude confrontation, the only difference is that in the experimental group a tree is presented near the participant whereas in the control group a parasol is presented at the same position. Thus the sentences that refer to the tree are changed in the audio of the control group. The height is increased to a maximum of 60 metres. Participants can stop the experiment at any time by pressing a button on a handheld joystick. During the confrontation, various events (e.g. rising balloons) generate additional altitude cues. The duration of the confrontation is approximately 15 minutes. Subsequently participants complete questionnaires about their fear of heights (HIQ) for a post-measurement of altitude anxiety and about their experience of presence (IPQ) and their experience of hypnotic depth (SSTT). Participants will undergo these questionnaires and the intervention three times within three weeks. On a separate day within these three weeks they will be placed in a 30-minute trance and given the Harvard Group Scale of Hypnotic Susceptibility (HGSHS) to test their suggestibility.

The total time required for the participants ist therefore approximately three hours and 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* HIQ-Score > 29
* informed consent

Exclusion Criteria:

* Negative previous experience with hypnosis
* Negative previous experience with virtual reality
* Mental illness (psychosis, post-traumatic stress disorder and/or personality disorder)
* neurological disease
* Acute or chronic disease (also anamnestic) that may affect brain metabolism:
* pre-existing diabetes mellitus (E10-E14 according to ICD-10)
* Renal insufficiency from stage 3 of the Kidney Disease Outcomes Quality Initiative
* Uncontrolled hypertension (I10.x according to ICD-10)
* Moderate or severe traumatic brain injury (GCS 3-12), or traumatic brain injury 2nd or 3rd degree with loss of consciousness of > 30 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Height intervention questionnaire (immediately before the intervention) | Immediately (circa 1 minute) before the height exposure in all three sessions
  Measurement of acrophobia
Height intervention questionnaire (immediately after the intervention) | Immediately (circa 1 minute) after the height exposure in all three sessions
  Measurement of acrophobia
Height intervention questionnaire (one-week-follow-up) | One week after the third height exposure
  Measurement of acrophobia
Height intervention questionnaire (three-months-follow-up) | Three months after the third height exposure
  Measurement of acrophobia
Subjective fear rating during height exposure | always 5 seconds after each rise in the height exposure in all three sessions
  Measurement of Fear on Likert scale (0 to 9)
Harvard Group Scale of Hypnotic Susceptibility (german brief form HGHSH-5) | at a separate day within the three weeks, where the interventions take place
  Measurement of Suggestibility (minimum value = 0, maximum value = 5, higher scores imply higher suggestibility)

SECONDARY OUTCOMES:
Subjective Scale for Trance Depth | (circa 5 minutes) after the height exposure in all three sessions
  Measurement of Trance Depth (minimum value = 38, maximum value = 152, higher scores imply higher subjective trance depth)
Igroup Presence Questionaire | (circa 3 minutes) after the height exposure in all three sessions
  Subjective Presence in the VR-experience (minimum value = -42, maximum value = +42, higher scores imply higher subjective presence)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Revenstorf, Prof., Principal Investigator — University Hospital Tuebingen
Locations (1):
- Department of Psychiatry and Psychotherapy, University Hospital Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
In the case of a publication of the results we will share deidentified individual participant data.
Supporting Information: SAP, Analytic Code
Time Frame: The data will become available when the results are published.

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT06618456/SAP_000.pdf